CLINICAL TRIAL: NCT07227467
Title: Prospective Assessments Following Immediate Lymphatic Reconstruction
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB25-1329
Record Dates: First submitted 2025-11-06; First posted 2025-11-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Lymphatic Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who are potential candidates for immediate lymphatic reconstruction (ILR): potential candidates for ILR based on possible nodal involvement assessed preoperatively.
  Interventions: Other: patients who are candidates for immediate lymphatic reconstruction

INTERVENTIONS:
Other: patients who are candidates for immediate lymphatic reconstruction — potential candidates for ILR based on possible nodal involvement assessed preoperatively.

SUMMARY:
Immediate lymphatic reconstruction (ILR) is a novel surgical approach performed at the time of initial lymph node dissection with the goal of preventing lymphedema.(Chang et al. 2020) It involves the identification of lymphatic channels that are transected after lymph node dissection and microsurgical anastomosis of one or more lymphatic channel with a local recipient vein to re-direct upper extremity lymphatic drainage. Although ILR carries significant promise in prevention of lymphedema, there is a lack of high-level evidence supporting its efficacy because it is a novel surgical technique that is only offered at a few centers and not routinely covered by insurance carriers yet. The University of Chicago Comprehensive Cancer Center (UCCCC) is one of the busiest microsurgery centers performing this procedure, and, as a Lymphedema Center of Excellence, is in a unique position to investigate the efficacy of ILR in preventing lymphedema. In addition, the University has access to a world class microbiome research facility and colleagues. To our knowledge, there is no information on the skin microbiome of the axilla in patients undergoing treatment for breast cancer or those at risk for developing lymphedema. Further exploratory studies such as this in a diverse patient population may lead to practice changing research in our approach to lymphedema management and prevention.

ELIGIBILITY:
Inclusion Criteria:

potential candidates for ILR based on possible nodal involvement assessed preoperatively.

Exclusion Criteria:

* Individuals who are not eligible for ILR based on possible nodal involvement assessed preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are potential candidates for ILR based on possible nodal involvement assessed preoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of immediate lymphatic reconstruction (ILR) based on limb circumference of each arm | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
the efficacy of immediate lymphatic reconstruction (ILR) based on volume | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
the efficacy of immediate lymphatic reconstruction (ILR) based on bioimpedance spectroscopy measurements of affected and unaffected limbs of women before and after surgery. | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
  Bioimpedance spectroscopy is a non-invasive technology that measures total body water, and both extracellular and intracellular fluid volumes.

SECONDARY OUTCOMES:
the impact of ILR on validated patient reported outcome tool using the lymphedema life impact scale (LLIS) | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
  This is an 18 questionnaire that has a scale from 0 (no pain) to 4 (severe pain)
the impact of ILR on validated patient reported outcome tool using The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
  This is a 30 questionnaire that has a scale from 1 (No difficulty) to 5 (unable)
the impact of ILR on validated patient reported outcome tool using the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
  This is a 10 questionnaire that scales from unable to do it (1) to not difficult (3).

OTHER OUTCOMES:
Comparison of the Axillary Microbiome in ILR-Treated and Untreated Limbs | post operative study period at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months and 60 months.
  Characterize the axillary microbiome in limbs that have been treated with ILR compared to those that were unaffected before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Hanson, MD, PhD, FACS, Principal Investigator — University of Chicago
Locations (1):
- The University o Chicago, Chicago, Illinois, United States